CLINICAL TRIAL: NCT06509035
Title: Correlation Between Smartphone Use and Text Neck Posture in Asymptomatic Subjects
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hend Hesham Abd Elfatah Ali, Principal Investigator, Cairo University
Other Study IDs: Hend PhD
Record Dates: First submitted 2024-07-02; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Smartphone Addiction; Text Neck Posture
Keywords: forward head posture; smart phone use
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will be conducted to investigate the correlation between the number of hours of smartphone usage and severity of text neck posture, cervical ROM, DNF endurance and resting head posture among asymptomatic 18 to 25 years old adults

DETAILED DESCRIPTION:
Smartphone use has increased significantly globally, with 79% of adults aged 18-44 carrying a smartphone constantly. This can cause excessive anterior curves in the neck vertebrae and increase the mechanical load on cervical spine joints. Overuse syndrome, spinal damage, and other side effects can result. This study aims to investigate the correlation between time spent using smartphones and text neck posture and its association with head and neck posture, cervical ROM, and DNF endurance among asymptomatic 18-25-year-olds.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who are willing to participate at the time of data collection.
2. Individuals aged 18 - 25 years old.
3. Individuals who use a smartphone to report the duration of weekly usage (at least one year of using a smartphone and minimum duration of smartphone use of ≥1 h per day

Exclusion Criteria:

1. Previous history of an accident or severe injury.
2. Any neurological or cardiovascular problem.
3. Spinal surgery or any disease that prevents the individual from adopting an unsupported orthostatic posture.
4. Congenital cervical problem.
5. Pregnant women.

Ages: 18 Years to 25 Years | Sex: All
Age Groups: Adult
Study Population: Thirty, males and females students, with age 18 - 25 years old recruited from faculty of physical therapy in Misr University for Science and Technology, 6 October, Egypt.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Assessing the average duration of smartphone screen time | at baseline
  A mobile application called Screen Time Restrain Yourself measures smartphone usage in hours over the past week, allowing users to monitor their daily usage without disrupting normal smartphone use.

SECONDARY OUTCOMES:
Assessment of head and neck posture | at baseline
  Photogrammetry is a reliable method for measuring head and cervical spine postures. It involves taking sagittal photographs of the subject's head tilt angle and neck tilt angle. A camera is positioned at a height corresponding to the seventh cervical vertebra (C7) level, and spherical markers are attached to the right tragus, canthus, and spinal process. The subject is instructed to sit on a chair, maintain a resting head posture, and perform full flexion and extension three times. The average of angles from repeated photos is used to reduce bias. Fatigue time is reported after ten minutes of use with a smartphone.
Assessment of cervical range of motion | at baseline
  Cervical ROM is measured using a universal goniometer, with subjects placed flat on the floor and supported on a lap. They move their head in flexion and extension, with the goniometer placed over the external auditory meatus, fixed arm perpendicular to the floor, and movable arm with the nose base. For cervical rotation, they turn the head to the left or right side, and for lateral flexion, they touch the ear to a shoulder of the same side. The goniometer is a valid and reliable tool for measuring cervical ROM, with good interrater and intraterrater reliability.
Assessment of deep neck flexor endurance | at baseline
  The Neck Flexor Muscle Endurance Test (NFMET) involves a subject supine, with hands resting on the abdomen and feet flat on a plinth. The subject performs chin retraction, head and neck lift, and skin folds. The test measures muscle endurance, with males having a longer average hold time than females.

CONTACTS AND LOCATIONS:
Locations (1):
- Misr University for Science and Technology, Giza, Egypt